CLINICAL TRIAL: NCT03903952
Title: Serum Levels of Folate And Vitamine B12 in Patients Infected With HPV and Diagnosed Atypical Squamous Cells of Undetermined Significance in Cervical Cytology
Brief Title: Can B12 and Folate Levels Predict HPV Penetration in Patients With ASCUS?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Collaborators: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nefise Nazlı YENIGUL, Ph.D. Assistant Professor Department of Obstetrics and Gynecology, Sanliurfa Mehmet Akif Inan Education and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 714
Record Dates: First submitted 2019-04-01; First posted 2019-04-04 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2014-05

CONDITIONS: ASC-US; Human Papilloma Virus
Keywords: ASCUS; HPV; Vitamine B12; Folate
MeSH Terms: conditions — Atypical Squamous Cells of the Cervix | interventions — Vitamin B 12; Folic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Papanicolaou smear result (control group) (Other): women who did not have intraepithelial neoplasia as a result of smear
  Interventions: Dietary Supplement: Vitamin B12 and folate
- Papanicolaou smear result (study group) (Other): women who have atypical squamous cells of undetermined significance (ASCUS) as a result of smear
  Interventions: Dietary Supplement: Vitamin B12 and folate

INTERVENTIONS:
Dietary Supplement: Vitamin B12 and folate — Vitamin B12 and folate levels in blood

SUMMARY:
Non-classified atypical squamous cells (ASCUS) is the most common abnormal cervical cytology (%39). The risk of cervical intraepithelial neoplasia 2-3 is 5% and the risk of carcinoma is around 0.1% after diagnosis. Mostly human papillomavirus (HPV) is responsible for this transition. Most of them are transient, but some infections become persistent and can progress into precancer and invasive cancer. In the process of progression to cancer; patients with cell cycle problems are thought to be at risk. In some studies, B12 and folate deficiency, which play a role in DNA synthesis and repair, have been shown to induce incorrect binding of uracil to DNA, leading to DNA breakage and repair disorder. Therefore, in this study, it has been aimed that the relation of presence of atypical squamous cells and HPV persistence with folate and vitamin B12 levels which effect on immune system.

DETAILED DESCRIPTION:
Participants were divided into two groups according to their smear results; atypical squamous cells of undetermined significance (ASCUS) (study group: 100 patients) and women who did not have intraepithelial neoplasia as a result of smear (control group: 100 patients). Patients who had well preserved sufficient number of squamous epithelial cells, who did not have bleeding, fixation failure, inflammation or atrophy, and had negative cervical cytology smear were considered as control group. HPV test was also requested from the study group. B12 and folate blood levels were compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* female patients aged between 30-65 who were undergoing smear tests with the aim of control
* body mass index (BMI) lower than 35
* Participants did not have any chronic diseases

Exclusion Criteria:

* Patients taking B12 and folate supplement due to mix type anemia
* patients taking active vitamin B12 and folate-containing vitamin supplements
* pregnant women
* women with other cervical intraepithelial lesions such as low grade squamous intraepithelial lesion (LGSIL), high grade squamous intraepithelial lesion (HGSIL) or high grade squamous intraepithelial lesion can not be excluded (ASC-H) in smear
* patients with cervical cancer diagnosis
* patients who were operated due to cervical cancer
* patients who had HPV vaccine
* patients with a diagnosis that can inhibit B12 and folate absorption in gastro-intestinal tract
* vegetarians

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2015-05-30 (Actual); Study Completion 2015-05-30 (Actual)

PRIMARY OUTCOMES:
the vitamine B12 levels . | 1 year
  the vitamine B12 levels in patients with ASCUS (+) smear.
The folate levels | 1 year
  the folate levels in patients with ASCUS (+) smear.